CLINICAL TRIAL: NCT00260442
Title: Egg Cholesterol Consumption, Blood Cholesterol and Skeletal Muscle Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Steven E.Riechman, PhD, MPH, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-0187; 481031-001-CA; 0600083
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia; Cardiovascular Disease
Keywords: sarcopenia; resistance training; strength training; skeletal muscle; elderly; cholesterol; aging; cardiovascular disease; nutrition; inflammation; lipids
MeSH Terms: conditions — Sarcopenia; Cardiovascular Diseases; Inflammation | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): < 200 mg/day dietary cholesterol, resistance training, sedentary
  Interventions: Behavioral: Resistance Training; Behavioral: Sedentary
- Average intake (Experimental): 400 mg/day dietary cholesterol, resistance training, sedentary
  Interventions: Behavioral: Resistance Training; Behavioral: Sedentary
- High intake (Experimental): 800 mg/day dietary cholesterol, resistance training, sedentary
  Interventions: Behavioral: Resistance Training; Behavioral: Sedentary

INTERVENTIONS:
Behavioral: Resistance Training — 12 weeks, 3 times a week whole body resistance training
Behavioral: Sedentary — Absence of physical activity

SUMMARY:
The purpose of this study is to examine the effect of dietary cholesterol administered as whole egg or egg white (control)on muscle mass gain with resistance training in a young old population of men and women (age 50-69). It is hypothesized that dietary cholesterol will be significantly associated to muscle mass gain.

DETAILED DESCRIPTION:
The primary objective of this proposal is to have 36 men and women (age 50-69) perform 12 weeks of resistance exercise training for the purpose of inducing skeletal muscle hypertrophy. These individuals will consume either 0, 1, or 3 whole eggs per day in a double-blind design to test the hypothesis that dietary cholesterol is essential for skeletal muscle hypertrophy. If so proven, this will confirm a very strong association between dietary cholesterol and hypertrophy observed in a previous study of 51 men and women (age 60-69). The current proposal is using a randomized double-blind, placebo controlled design to provide the most conclusive evidence that dietary cholesterol plays an essential role in skeletal muscle hypertrophy.

The secondary objective of this proposal is to test the hypothesis that increased dietary cholesterol consumption in the context of an exercise program does not alter blood cholesterol concentrations or other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 50-69
* able to perform exercise testing and training

Exclusion Criteria:

* blood pressure > 160/100
* cardiac arrhythmias
* cancer
* hernia
* aortic aneurysm
* kidney disease
* lung disease
* total cholesterol > 240 mg/dl or < 160 mg/dl
* current use of cholesterol lowering medications
* actively participating in >1 hour per week of resistance training

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Primary: Strength and muscle gain (DEXA) | after 12 weeks of resistance training

SECONDARY OUTCOMES:
Secondary: Blood lipids, inflammatory markers, blood pressure | after 12 weeks of resistance training

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Riechman, PhD, MPH, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States